CLINICAL TRIAL: NCT06186388
Title: TEMPO (iMOvifa) Glaucoma Screening
Brief Title: Glaucoma Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cape Fear Eye Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CF-2023-01
Record Dates: First submitted 2023-12-15; First posted 2024-01-02 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Pathology (Other): Subjects with glaucoma-affected eyes
  Interventions: Diagnostic Test: TEMPO iMOvifa
- Normal (Other): Subjects with healthy eyes
  Interventions: Diagnostic Test: TEMPO iMOvifa

INTERVENTIONS:
Diagnostic Test: TEMPO iMOvifa — Screening test with 28 testing points

SUMMARY:
* The primary objective of this study is to evaluate the diagnostic accuracy of the TEMPO (iMOvifa) visual field perimeter screening test by measuring the sensitivity in a population of eyes with glaucoma and the specificity in a population of normal eyes and to measure repeatability of the screening test.
* The secondary objective of this study is to gather and analyze ancillary data to confirm the diagnosis or absence of glaucoma.

ELIGIBILITY:
Inclusion Criteria (All subjects):

* Subjects 40 years of age or older on the date of informed consent.
* Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent.
* BCVA 20/40 or better in both eyes.

Inclusion Criteria- Normal Population

* IOP ≤ 21 mmHg
* Healthy anterior and posterior segment evaluation on clinical examination.

Inclusion Criteria - Pathology Population

• Diagnosis of glaucoma on clinical examination.

Exclusion Criteria (All subjects):

* Unable to tolerate ophthalmic imaging and/or diagnostic testing.
* History of intraocular surgery (uncomplicated surgeries are accepted).
* Ocular diseases including uveitis, non-glaucomatous optic neuropathy, severe or proliferative diabetic/ hypertensive retinopathy (controlled diabetes and hypertension participants with no or mild to moderate retinopathy [not involving the macula] can be included), unresolved trauma.
* Any neurodegenerative diseases including Alzheimer, Parkinson, or dementia, or history of stroke.
* Unreliable VF testing and/or poor-quality OCT scans.
* Poor fixation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity | 1 day
  sensitivity in a population of eyes with glaucoma and specificity in a population of normal eyes

SECONDARY OUTCOMES:
RNFL and GCL thickness | 1 day
  Using Maestro2 OCT

CONTACTS AND LOCATIONS:
Overall Officials: Christina Jones, Study Director — Clinical Research Coordinator
Locations (1):
- Cape Fear Eye Institute, Wilmington, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No